CLINICAL TRIAL: NCT06838949
Title: A Clinical Study on the Efficacy and Safety of Herombopag in the Treatment of Senile Primary Immune Thrombocytopenia
Brief Title: A Clinical Study on the Efficacy and Safety of Herombopag in the Treatment of Senile Primary ITP
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2023054
Record Dates: First submitted 2025-01-21; First posted 2025-02-21 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-01

CONDITIONS: Herombopag

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Herombopag (Experimental): Herombopag 2.5mg per tablet
  Interventions: Drug: herombopag olamine tablets

INTERVENTIONS:
Drug: herombopag olamine tablets — The patient received herombopag 5mg/d at the beginning of the day, was orally taken on an empty stomach in the morning, and could eat 2 hours after taking the drug, once a day for 24 weeks. Investigators will adjust the dosage of herombopag once a week according to the platelet count, with a maximum dosage of 7.5 mg per day. Efficacy and safety were evaluated once a week.

SUMMARY:
The objective of this study was to evaluate the efficacy and safety of Herombopag in the treatment of elderly patients with ITP.

DETAILED DESCRIPTION:
This is a single-arm, prospective clinical study to evaluate the efficacy and safety of herombopag in the treatment of elderly patients with ITP. The study will include 80 patients. Screening of patients will be 2 weeks after the longest period, to enter after the treatment period, accept the herombopag 5 mg, once daily, on an empty stomach, oral medication can be eating only 2 hours, and 24 weeks of treatment, and adjust the dosage according to the platelet count. If patients do not respond to treatment after 8 weeks, it is recommended to withdraw from the study and continue safety visits for 4 weeks. During treatment, the patient continues treatment until the investigator assesses the occurrence of intolerable toxicity, disease progression, withdrawal of informed consent, or other discontinuation criteria specified in the protocol (whichever occurs first). Follow-up treatment for patients who withdraw from treatment due to safety or ineffectiveness is determined by the investigator according to clinical practice. Safety assessment during treatment, including vital signs, physical examination, laboratory examination, etc.; Check your blood routine at least once a week. A 4-week safety visit was performed after the final treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients voluntarily participated in the study and signed informed consent;
* Age ≥60 years old, gender unlimited;
* ECOG PS ≤2;
* Expected survival ≥6 months;
* A definitive diagnosis of ITP, including newly diagnosed, chronic, and persistent ITP;
* PLT < 30×109/L for at least two consecutive times with an interval of at least 1 day before medication
* Patients with laboratory test results meet the following criteria: a. alanine aminotransferase (ALT) 3.0 x or less normal limit (ULN), aspartate aminotransferase (AST) 3.0 x ULN or less; b. Serum total bilirubin ≤1.5×ULN; c. Serum creatinine ≤1.5×ULN;
* The researchers determined that patients could be treated with hexapopal.

Exclusion Criteria:

* Patients who did not respond to previous treatment with herombopag;
* A history of allergy to thrombopoietin receptor agonist (TPO-RA) drugs;
* Combined with other important organ dysfunction, such as liver and kidney failure, cardiac insufficiency, etc.
* Secondary thrombocytopenia, such as rheumatic immune disease, chronic liver disease, hyperlienism, malignant hematologic disease, bone marrow hematopoietic exhaustion disease (such as AA, MDS), hereditary thrombocytopenia, CVID, drug-induced thrombocytopenia, etc.;
* Receive TPO-RA medication within 2 weeks prior to treatment;
* Non-steroidal anti-inflammatory drugs (aspirin, salicylate, etc.) and anticoagulants (warfarin, clopidogrel, etc.) should be taken during treatment, which have an impact on platelet function.
* There are severe active bleeding symptoms, such as gastrointestinal bleeding, intracranial bleeding, etc.
* Severe thrombotic disease, such as transient ischemic attack, myocardial infarction, pulmonary embolism, deep vein thrombosis, and disseminated intravascular coagulation (DIC), occurred within 6 months prior to the screening period;
* Have a New York Heart Society (NYHA) Class 3 or 4 congestive heart failure, or have a history of NYHA Class 3/4 congestive heart failure with a left ejection fraction (LVEF) of < 45% within 4 weeks prior to treatment;
* Positive anti-human immunodeficiency virus antibody or anti-treponema pallidum specific antibody; Hepatitis virus positive, such as HBV, HCV, etc.
* A history of cirrhosis;
* Bone marrow reticulum fiber staining (MF) ≥2 grade;
* Have an active infection that is difficult to control;
* Have a history of or accompanied by malignant tumors;
* Pregnant or lactating women;
* Any other conditions that the investigator determines are not suitable for participation in the study.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-03-03 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with platelet count ≥30×109/L | 8 weeks
  Proportion of subjects with a platelet count ≥ 30 × 10^9/L and at least twice the baseline platelet count without bleeding at week 8

SECONDARY OUTCOMES:
Proportion of patients with platelet count ≥50×109/L | 8 weeks
  Proportion of patients with platelet count ≥50×109/L within 8 weeks of treatment
Proportion of patients with platelet count ≥100×109/L | 8 weeks
  Proportion of patients who achieved CR within 8 weeks of treatment
Duration from treatment initiation to platelet count ≥30×10^9/L and ≥50×10^9/L | 24 weeks
  The time of first Platelet≥30×109/L and ≥50×109/L
Sustained response at 24 weeks of treatment | 24 weeks
  Sustained response at 24 weeks of treatment defined as 8 weeks after the last visit, at least 6 visits with platelets ≥30×109/L, greater than 2 times of baseline, and no bleeding
The change in bleeding score before treatment and 8 weeks after treatment assessed using the world health organization (WHO) bleeding scale | 8 weeks
  The change in bleeding score before treatment and 8 weeks after treatment according to the reported World Health Organization's Bleeding Scale. The WHO Bleeding Scale is a measure of bleeding severity with the following grades: grade 0 = no bleeding, grade 1= petechiae, grade 2= mild blood loss, grade 3 = gross blood loss, and grade 4 = debilitating blood loss.
Emergency treatment | 8 weeks
  The proportion of subjects who received emergency treatment within 8 weeks and during the entire study period.
incidence of treatment-emergent Adverse Events and TRAE | 24 weeks
  Incidence, severity, and relationship of treatment emergent adverse events after treatment as assessed by CTCAE v5.0

CONTACTS AND LOCATIONS:
Overall Officials: Yunfei Chen, Principal Investigator — Chinese Academy of Medical Science and Blood Disease Hospital
Locations (1):
- Chinese academy of medical science and blood disease hospital, Tianjin, China

IPD SHARING:
Plan to Share IPD: No